CLINICAL TRIAL: NCT04684550
Title: Randomized Controlled Clinical Study (RCT) Phase 3 of the Safety and Efficacy of Hypochlorous Acid in the Prophylaxis of Healthcare Personnel at High Risk of Infection by SARS-CoV2 (COVID19) Versus Placebo
Brief Title: Use of Hypochlorous Acid as Prophylaxis in Health Personnel at High Risk of Infection by SARS-CoV 2 (COVID19)
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study did not achieve funding or approval by the ethics committee. Once the vaccination phase was entered, the study lost validity and was not viable
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FM-CIE-0824-20
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV Infection; Covid19; Infection Viral
Keywords: SARS-CoV Infection; Stabilized hypochlorous acid (S-HClO); Prophylaxis; Health Professionals
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Virus Diseases

STUDY DESIGN:
Intervention Model Description: A randomized, double-masked, placebo-controlled clinical experiment is proposed.
Who Masked: Participant, Care Provider, Investigator
Masking Description: * The first group of health personnel who work in places of greater risk (hospitals and primary level consultation) with conventional protection elements added to the application of 2 nasal puff every 8 hours of a nasal spray containing 0.9% SSN (placebo) and gargles (SSN 0.9%).
  * A second group of health personnel who work in higher risk places (hospitals and primary level consultation) with conventional protection elements added to the application of 2 puffs and gargles every 8 hours of a solution with low concentrations of S-HCLO (3-5 ppm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Health personnel who work in places of greater risk (hospitals and primary level consultation) with conventional protection elements added to the application of 2 nasal puff every 8 hours of a nasal spray containing 0.9% SSN (placebo) and gargles (SSN 0.9%).
  Interventions: Drug: Placebo
- Experimental (Experimental): Health personnel who work in higher risk places (hospitals and primary level consultation) with conventional protection elements added to the application of 2 puffs and gargles every 8 hours of a solution with low concentrations of S-HCLO (3-5 ppm).
  Interventions: Drug: Stabilized hypochlorous acid

INTERVENTIONS:
Drug: Stabilized hypochlorous acid — Application of 2 puffs and gargles every 8 hours of a solution with low concentrations of S-HCLO (3-5 ppm).
  Arms: Experimental
Drug: Placebo — Application of 2 puffs and gargles every 8 hours of a solution with low concentrations of S-HCLO (3-5 ppm).
  Arms: Placebo

SUMMARY:
The pandemic caused by SARS-CoV-2 is a global emergency present in 6 continents including 66 countries, incurring a shortage of effective and safe therapeutic alternatives that can contribute to reducing the risk of contamination, as well as helping to reduce the viral load of the positive patient. This requires a coordinated, effective and immediate action on the part of governments, companies, academic entities and even at the individual level.

In the search for new therapeutic and prevention alternatives, the application of hypochlorous acid (HClO) to the nasal mucosa is proposed, a broad-spectrum and fast-acting antimicrobial solution, whose safety has been proven in preclinical trials. The efficacy of HClO has been tested against enveloped and non-enveloped viruses, reducing virus particles without affecting human cells. This solution could contribute to reducing the viral load and the risk of contamination of patients and professionals. This could have an impact on controlling the COVID-19 pandemic.

DETAILED DESCRIPTION:
Hypochlorous acid (HClO) is a powerful antimicrobial and antiviral used for the control of various infections, repair and washing of surgical wounds, as well as for disinfection of surfaces. In vivo, it is synthesized by the cells of the immune system for the control of pathogens during phagocytosis and has been synthesized and stabilized for use in different entities.

The therapeutic uses of HClO began in the First World War with the studies of Alexis Carrel and Henry Dakin who obtained a buffered sodium hypochlorite solution (Dakin's solution) which generated ideal concentrations of HClO, using it successfully in washing and treatment of wounds without presenting any damage or undesired effect on the patient's tissues. In 1993, the HClO molecule was stabilized, popularizing its use for the control of predominantly skin infections, treatment of chronic ulcers, closure and cleaning of wounds, management of burned patients, and disinfection of surfaces.

Biologically, it is part of the reactive oxygen species (ROS) synthesized by cells of the immune system (Neutrophils and Macrophages) during an immunological process known as "respiratory burst", during phagocytosis of antigens in reaction with the enzyme myeloperoxidase (MPO), hydrogen peroxide (H2O2) and a chlorine ion. Safety profiles in in vivo models have driven our initiative to use Stabilized Hypochlorous Acid (S-HClO), as an early therapeutic option in patients with SARS-Cov-2 infection or in close contact with COVID-193 positive patients.

Calderon et al and carried out the evaluation of the antimicrobial effect of HClO on potentially pathogenic microorganisms of the oral cavity. The study reports that hypochlorous acid achieved bacterial inhibition of 99.9% at a concentration of 0.05% and a pH of 5.2 per minute of action for different types of bacteria and for infectious microorganisms. Virological tests have also been performed on feline calcivirus (Ebola-like virus), rotavirus, AH1N1, adenovirus and SARS, found to be highly effective after 1 minute of application.

In the face of the COVID-19 pandemic, effective and early treatments are being sought to help prevent the dissipation of the virus (disinfection of surfaces), to neutralize the virus at an early stage when it is lodged in the upper respiratory tract and nose, since this is the Probable route of infection of the ethmoid lamina and later causing viral encephalopathy and treatment of patients with bronchial infection by this virus, decreasing the viral load and causing destruction of the virus. There are reports of the use of HClO in the nasal mucosa in studies in humans, reporting safety and effectiveness, both in adults and in children, which leads us to propose the application of said nasal spray solution, as a prophylaxis in health personnel with a high risk of infection by SARS-CoV-2.

A RCT with the use S-HClO as a prevention treatment for the infection by SARS-CoV-2 in health professionals is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Specialist physicians, resident physicians, medical students, and nursing personnel who work at the San Ignacio University Hospital.
* Subjects of any sex over 18 years of age who work as health care personnel, in care services that care for patients with a suspected or confirmed diagnosis of COVID-19 and who are active during the study recruitment.
* That they have not presented general symptoms such as malaise, fever, cough, dyspnea or muscle pain during the last 7 days.
* Subjects negative to the antigen test for COVID-19.

Exclusion Criteria:

* Subjects considered as a resolved case of COVID-19 infection, according to guidelines from the Colombian National Institute of Health.
* Health personnel with social distancing due to close contact without personal protective equipment with patients confirmed to be infected or taking any medication as a possible prophylaxis for COVID-19 (example: chloroquine, hydroxychloroquine, azithromycin)
* Health workers who have permits or temporary withdrawal from their hospital work for more than one week during the month of the study.
* Some type of allergy to chlorinated agents or hypersensitivity to HClO
* Known diagnosis of upper airway respiratory disease where COVID-19 such as the common cold, sinusitis, pharyngitis, laryngotracheitis and epiglottitis or lower such as bronchiolitis, pneumonia, and mixed conditions have been ruled out.
* Previous COVID19 infection determined by positive PCR or positive serum antibody titers.
* Any condition that in the principal investigator's discretion renders the subject ineligible to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Prevention of infection by COVID19 | Through study completion, an average of 6 months
  Number of participants who get COVID19 infection during the application of S-HClO

SECONDARY OUTCOMES:
Adverse drug reaction (ADR) | Through study completion, an average of 6 months
  Determine the occurrence of ADR by the use of S-HClO
Seroconversion | Through study completion, an average of 6 months
  Determine the frequency of seroconversion due to COVID 19
Hospitalization | Through study completion, an average of 6 months
  Number of participants who fell ill from COVID-19 and was not hospitalized
ICU | Through study completion, an average of 6 months
  Number of participants who fell ill from COVID-19 and was hospitalized in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Juan Zambrano, MD. M.Sc., Principal Investigator — Hospital Universitario San Ignacio/Pontificia Universidad Javeriana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hui DS, Chan PK. Severe acute respiratory syndrome and coronavirus. Infect Dis Clin North Am. 2010 Sep;24(3):619-38. doi: 10.1016/j.idc.2010.04.009. PMID 20674795
- [Background] Velavan TP, Meyer CG. The COVID-19 epidemic. Trop Med Int Health. 2020 Mar;25(3):278-280. doi: 10.1111/tmi.13383. Epub 2020 Feb 16. No abstract available. PMID 32052514
- [Background] Gold MH, Andriessen A, Bhatia AC, Bitter P Jr, Chilukuri S, Cohen JL, Robb CW. Topical stabilized hypochlorous acid: The future gold standard for wound care and scar management in dermatologic and plastic surgery procedures. J Cosmet Dermatol. 2020 Feb;19(2):270-277. doi: 10.1111/jocd.13280. Epub 2020 Jan 6. PMID 31904191
- [Background] Hakim H, Thammakarn C, Suguro A, Ishida Y, Kawamura A, Tamura M, Satoh K, Tsujimura M, Hasegawa T, Takehara K. Evaluation of sprayed hypochlorous acid solutions for their virucidal activity against avian influenza virus through in vitro experiments. J Vet Med Sci. 2015 Feb;77(2):211-5. doi: 10.1292/jvms.14-0413. Epub 2014 Nov 24. PMID 25421399
- [Background] Taharaguchi M, Takimoto K, Zamoto-Niikura A, Yamada YK. Effect of weak acid hypochlorous solution on selected viruses and bacteria of laboratory rodents. Exp Anim. 2014;63(2):141-7. doi: 10.1538/expanim.63.141. PMID 24770639
- [Background] Ishihara M, Murakami K, Fukuda K, Nakamura S, Kuwabara M, Hattori H, Fujita M, Kiyosawa T, Yokoe H. Stability of Weakly Acidic Hypochlorous Acid Solution with Microbicidal Activity. Biocontrol Sci. 2017;22(4):223-227. doi: 10.4265/bio.22.223. PMID 29279579
- [Background] Edward DG, Lidwell OM. Studies on air-borne virus infections: III. The killing of aerial suspensions of influenza virus by hypochlorous acid. J Hyg (Lond). 1943 Sep;43(3):196-200. doi: 10.1017/s002217240001281x. No abstract available. PMID 20475674
- [Background] Yu MS, Kim BH, Kang SH, Lim DJ. Low-concentration hypochlorous acid nasal irrigation for chronic sinonasal symptoms: a prospective randomized placebo-controlled study. Eur Arch Otorhinolaryngol. 2017 Mar;274(3):1527-1533. doi: 10.1007/s00405-016-4387-5. Epub 2016 Nov 17. PMID 27853946